CLINICAL TRIAL: NCT02966925
Title: Evaluation of the Benefit of the Use of Platelet-Rich Plasma (PRP) Combined to Hyaluronic Acid (HA) for Vulvovaginal Dryness
Brief Title: Autologous Platelet Concentrate Combined to Hyaluronic Acid Obtained With Cellular Matrix® BCT-HA Kit and Vulvovaginal Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regen Lab SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-SM-001
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Vulvar Atrophy
Keywords: Vulvovaginal dryness

STUDY DESIGN:
Intervention Model Description: case-series
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Cellular Matrix (Experimental): Patients will be treated with a combination of PRP/HA prepared with Cellular Matrix BCT-HA Kit
  Interventions: Device: Cellular Matrix BCT-HA Kit

INTERVENTIONS:
Device: Cellular Matrix BCT-HA Kit — Submucosal injections in the vulva, in the posterior vaginal wall and in the perineum of a combination product made of PRP and HA prepared using the Cellular Matrix BCT-HA medical device

SUMMARY:
Vulvovaginal irritation is a frequent complaint among postmenopausal women. Common symptoms of vaginal atrophy include dryness, itching, burning and dyspareunia.

This pilot study will assess the efficacy of platelet-rich plasma (PRP) combined to hyaluronic acid (HA) to relieve vulvovaginal dryness in patients who cannot benefit from reference treatments (hormonal therapies).To achieve this, 20 patients suffering from vulvovaginal dryness will be treated with one session of injections in the vulva, the posterior vaginal wall and the perineum, and followed-up for 6 months. Improvement of vaginal dryness will be primarily appreciated through Friedmann score and pH value, and secondarily through the Female Sexual Function Index (FSFI), as measured at baseline and 1, 3 and 6 months after the treatment.

DETAILED DESCRIPTION:
A treatment relying on the association of both platelet-rich plasma (PRP) and hyaluronic acid (HA) could represent a therapeutical alternative for patients suffering from vulvovaginal dryness who cannot be treated with hormone therapy.

Indeed, hyaluronic acid is widely distributed in all tissues, and most particularly in vulvovaginal tissues. Due to its hydrating and healing properties, HA plays a key role in tissue regeneration, facilitating the entry of a large number and variety of cells into the injured area, reconstructing in this way an extracellular matrix capable of supporting the proliferation and differentiation of cells for tissue regeneration. In addition,its ability to retain water at up to 1000x its weight makes it the ideal substance for ensuring hydration of the skin. Thus, the gynaecological use of HA could be a promising therapeutic option for the treatment of vulvovaginal dryness.

On the other hand, numerous studies have shown the role of PRP in the healing of soft and hard tissues. PRP is an autologous preparation from the patient's own blood playing the role of growth factors reservoir during treatment. Indeed, platelet activation induces alpha-granules degranulation, releasing synthesized pre-packaged growth factors. Once released, growth factors induce different cell signaling cascades that activate angiogenesis, cell proliferation, cell differentiation and new matrix synthesis for tissue regeneration. A recent clinical study showed that PRP could significantly reduce sexual distress of patients suffering from dyspareunia and suggests that PRP could improve vaginal vascularization and physiologic responsivness in patients with vaginal atrophy.

In the present pilot study, a combination of PRP/HA obtained with Cellular Matrix will be injected in the vulva, vaginal wall and perineum of women with vulvovaginal dryness. Outcomes will be compared before and at various timepoints after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from vulvovaginal dryness who cannot benefit from hormonal therapy
* Patients having signed an Informed Consent
* Patient capable of understanding the study's imperatives

Exclusion Criteria:

* Vulvovaginal inflammation or infection
* History of vaginal herpes
* History of vulvar, vaginal or cervical cancer
* Lichen sclerosus
* History of allergy to HA
* Hereditary or acquired hematological or clotting disorders, such as drepanocytosis, platelet dysfunction, thrombocytopenia (150'000 platelets/µl)
* Anemia (HGB ≤ 10g/dl)
* Autoimmune disease (Hashimoto, rheumatoid disease, lupus, etc.)
* HIV positive
* Hepatitis B or C
* Pregnancy or breastfeeding
* No contraception

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Vaginal pH | 3 months
  Variation of the vaginal pH between baseline and Month 3 after treatment
Friedmann score | 3 months
  Variation of the Friedmann score between baseline and Month 3 after treatment

SECONDARY OUTCOMES:
Female Sexual Distress (FSD) score | Month 1, Month 3 and Month 6
  Variation of the FSD score between baseline and various timepoints after treatment
Female Sexual Function Index (FSFI) score | Month 1, Month 3 and Month 6
  Variation of the FSFI score between baseline and various timepoints after treatment
Adverse device effects | Month 1, Month 3 and Month 6
  Safety monitoring through the record of adverse device effects at Month 1, Month 3 and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Méningaud, MD, Principal Investigator — CHU Henri Mondor
Locations (1):
- Centre Hospitalier Universitaire Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No